CLINICAL TRIAL: NCT03257696
Title: Diagnostic Accuracy Study of an Answer Reliability Assessment Tool for Aphasic Patients
Brief Title: Yes/No Questionnaire for Aphasic Patients (YNQ)
Acronym: YNQ
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/P03/031
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Stroke, Acute; Aphasia
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Close-ended questionnaire — Yes/no questionnaire used in order to identify "reliable respondent" and "unreliable respondent"

SUMMARY:
Quality of care depends strongly on oral communication with patients. Stroke patients, who have language disorders, have understanding difficulties, but also have difficulties in expressing their needs and in being understood. Available tools do not allow a professional consensus on the assessment of patients' ability to answer reliably to questions asked by caregivers. The investigators propose an answer reliability assessment tool based on yes or no questions. The goal of the present study is to define an optimal score for defining the test positivity, as a compromise between sensitivity and specificity, and by emphasizing the negative predictive value.

DETAILED DESCRIPTION:
In France, about 130,000 persons per year are victims of stroke. Thirty percent of the victims suffer from aphasia during the acute phase. These language impairments have an impact on caregiving. In the context of post-stroke aphasia, the most relevant means of verbal communication is closed-ended questioning. However, the available tools do not allow a professional consensus and the comprehensive assessment tools for aphasia do not provide any indication of the reliability of patients' answers. The investigators have developed a tool, the yes/no questionnaire that consists of 10 closed-ended questions designed to assess the patient's ability to provide a coherent answer. During one year, successive patients taken care in the neurovascular unit at la Rochelle hospital will be assessed for eligibility to the study and their relative will be informed and ask for consent. Aphasic patients will therefore answer the yes/no questionnaire. Based on the speech therapist evaluation, patients will be classified as "reliable respondent" or "unreliable respondent".

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Left-sided stroke
* Right-handed
* Mother language: French
* Hospitalized in neurovascular unit or neurology department
* NIHSS score over 25

Exclusion Criteria:

* Deaf
* Psychiatric history
* Stroke history
* Dementia or pre-stroke cognitive impairment
* Under guardianship
* Refusal to participate (relatives)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Right-handed, adult patients who are taken care in the neurovascular unit and in the neurology department because of a left stroke
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélia RAVIER-CUETO, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Reliable: Patients who respond reliably to closed questions, according to the speech therapist classification
- Unreliable: Patients who do not respond reliably to closed questions, according to the speech therapist classification
Period: Overall Study
Arm/Group | Reliable | Unreliable
Started | 123 | 29
Completed | 123 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reliable | Unreliable | Total
Number analyzed (Participants) | 123 | 29 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 7 | 32
  >=65 years | 98 | 22 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (12.8) | 75.4 (14.7) | 72.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 17 | 74
  Male | 66 | 12 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 123 | 29 | 152
Diagnostic [Count of Participants; unit: Participants]
  Ischemic stroke | 109 | 24 | 133
  Hemorrhagic stroke | 11 | 4 | 15
  Combination of both stroke subtypes | 3 | 1 | 4
Thrombolysis [Count of Participants; unit: Participants]
  Thrombolysis | 29 | 6 | 35
  No thrombolysis | 94 | 23 | 117

OUTCOME MEASURES:

1. Primary Outcome: YNQ Score
Description: The Yes/No questionnaire consists in 10 closed-ended questions designed to assess the patient's ability to provide a coherent answer.
  It was designed with questions that are very easy to answer, with the following constraints:
  * The questionnaire use only the auditory/verbal channel .
  * The questions ask only about personal data because they are less ambiguous.
  * The syntactical construction of the questions is very simple.
  * Apart from the use of personal data very familiar to the participants, the other nouns in the closed questions are very frequent (according to a lexical database).
  * The length of the questions was limited to seven words.
  * With the exception of two questions, each yes-response question had a no-response equivalent, as in some existing tests.
  A score of zero indicates a wrong answer to all questions. A score of ten indicates a correct answer to all questions.
Time Frame: measured within 7 in-hospital days
Measure: Count of Participants; unit: Participants
Arm/Group | Reliable | Unreliable
Number analyzed (Participants) | 123 | 29
Participants
  YNQ score = 0 | 0 | 1
  YNQ score = 1 | 0 | 1
  YNQ score = 2 | 0 | 0
  YNQ score = 3 | 0 | 2
  YNQ score = 4 | 1 | 1
  YNQ score = 5 | 0 | 4
  YNQ score = 6 | 0 | 4
  YNQ score = 7 | 1 | 5
  YNQ score = 8 | 0 | 4
  YNQ score = 9 | 0 | 2
  YNQ score = 10 | 121 | 5

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Reliable | Unreliable
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/29
Other Adverse Events (participants affected / at risk) | 0/123 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT03257696/Prot_SAP_000.pdf